CLINICAL TRIAL: NCT03932773
Title: Multi-site Confirmatory Efficacy Treatment Trial of Combat-related PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Collaborators: University of Texas Southwestern Medical Center (Other); Johns Hopkins University (Other); Metrocare Services of Dallas (Unknown); Florida State University (Other)
Responsible Party: Principal Investigator, John Hart, Jr., Professor, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-123; CDMRP-BA160594 (Other Grant/Funding Number: CDMRP)
Record Dates: First submitted 2019-04-04; First posted 2019-05-01 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PTSD; post-traumatic stress disorder; military-related PTSD; CPT; cognitive processing therapy; rTMS; repetitive transcranial magnetic stimulation; combat; combat-related PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three treatment arms: (1) 1 Hz (hertz) repetitive transcranial magnetic stimulation (rTMS) to the right dorsolateral prefrontal cortex (rDLPFC) coupled with Cognitive Processing Therapy (CPT), (2) sham rTMS coupled with CPT, or (3) 1 Hz rTMS to the rDLPFC alone.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Cognitive Processing Therapists will be blind to the treatment arm to which the participants are assigned.
  Baseline and outcome measure neuropsychological assessments will be conducted by an independent, blinded evaluator who is not part of the treatment team.
  Electroencephalography and magnetic resonance imaging data will be collected by technicians who are blinded to the arm to which the participants are assigned.
  Technicians administering repetitive transcranial magnetic stimulation (rTMS) will be blind to whether they are using an active or sham coil and to the treatment arm to which the participants are assigned. The coils are identical and will be setup by a different technician.
  Participants assigned to the 1 Hz rTMS coupled with Cognitive Processing Therapy or sham rTMS coupled with CPT will be blind as to whether they are receiving active or sham rTMS.
  Participants receiving rTMS only will not be blind to their group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Sham rTMS + CPT (Sham Comparator): 30 minutes of sham repetitive transcranial magnetic stimulation (rTMS) to the right dorsolateral prefrontal cortex (rDLPFC) prior to each Cognitive Processing Therapy (CPT) session
  Interventions: Device: Active rTMS; Behavioral: Cognitive Processing Therapy
- Active rTMS + CPT (Active Comparator): 30 minutes of 1 Hz rTMS to rDLPFC prior to each CPT session
  Interventions: Device: Sham rTMS; Behavioral: Cognitive Processing Therapy
- Active rTMS Alone (Active Comparator): 30 minutes of 1 Hz rTMS to rDLPFC at 1 session per week over 12 weeks
  Interventions: Device: Active rTMS

INTERVENTIONS:
Device: Active rTMS — A Magstim Rapid2 Stimulator repetitive transcranial magnetic stimulation (rTMS) device will be used to deliver 1 hertz (Hz) stimulation to right dorsolateral prefrontal cortex (rDLPFC) at 110% of a participant's rTMS motor threshold. The device passes electric current through a coil generating an alternating magnetic field. When positioned over the skull, the changing magnetic field causes electromagnetic inducted current flow in brain regions subjacent to the coil. Magnetic pulses (1.5-2.0 Tesla) lasting 100-300 microseconds at 1 Hz will be used.
  Motor threshold will be defined by the TMS intensity to right motor region required to induce visually perceptible movement of the contralateral abductor pollicus brevis 50 percent of the time.
  Other Names: 1 Hz repetitive transcranial magnetic stimulation
  Arms: Active rTMS Alone; Sham rTMS + CPT
Device: Sham rTMS — A Magstim Rapid2 Stimulator repetitive transcranial magnetic stimulation (rTMS) device will be paired with sham coil. The sham coil will induce electrical current flow in the tissue above the skull but will not induce current flow in brain tissue. The sham coil will be placed over the right prefrontal scalp region to target current flow in rDLPFC. Magnetic pulses lasting for 100-300 microseconds at 1 Hz will be used.
  For consistency across the rTMS conditions, motor threshold in the sham condition also will be determined by positioning the active rTMS coil over the right motor region and identifying the stimulation intensity required to induce visually perceptible movement of the contralateral abductor pollicus brevis 50 percent of the time.
  Other Names: sham repetitive transcranial magnetic stimulation
  Arms: Active rTMS + CPT
Behavioral: Cognitive Processing Therapy — Cognitive Processing Therapy (CPT) is an evidenced based, trauma-focused treatment for Posttraumatic Stress Disorder (PTSD). CPT is a recommended form of treatment in the Veterans Administration - Department of Defense Clinical Practice Guideline for PTSD. The CPT manual delineates the agenda for each of 12 sessions (60 minutes per session): 1) Introduction to CPT and Patient Education regarding PTSD, 2) Meaning of the Trauma, 3) Identification of Thoughts and Feelings related to the Trauma, 4) Remembering the Trauma, 5) Identification of Stuck points, 6) Challenging Questions about the Trauma, 7) Dysfunctional/Maladaptive Thinking patterns related to the Trauma, 8) Safety Issues, 9) Trust Issues, 10) Power and Control Issues, 11) Self-Esteem Issues, and 12) Intimacy Issues.
  Other Names: CPT
  Arms: Active rTMS + CPT; Sham rTMS + CPT

SUMMARY:
The purpose of this study is to examine the benefits of combining repetitive Transcranial Magnetic Stimulation (rTMS) coupled with Cognitive Processing Therapy (CPT) in treating combat-related Posttraumatic Stress Disorder (PTSD) symptoms. The study will also examine change in depression, psychosocial functioning, and neurophysiological (i.e., electroencephalography and magnetic resonance images) measures.

DETAILED DESCRIPTION:
Using three treatment arms, the study will examine Posttraumatic Stress Disorder (PTSD) symptom reduction when (1) 1 Hz (hertz) repetitive transcranial magnetic stimulation (rTMS) to the right dorsolateral prefrontal cortex (rDLPFC) is administered prior to each of 12 Cognitive Processing Therapy (CPT) sessions compared to when (2) sham rTMS is administered to the rDLPFC is administered prior to each of 12 CPT sessions and to when (3) 1 Hz rTMS is delivered to rDLPFC alone over 12 sessions.

Veterans with combat-related PTSD will be randomly assigned to one of the three treatment arms. Primary outcome PTSD symptom severity measures, secondary neuropsychological, electroencephalography (EEG), and magnetic resonance imaging (MRI) outcome measures, and prescreening assessments for study contraindicators will be collected prior to being assigned to a treatment arm (i.e., baseline).

Primary outcome PTSD symptom severity measures and secondary neuropsychological outcome measures will be collected twice within the span of the treatment sessions (i.e., sessions 5 and 9) and at three times following treatment competition (i.e., 1-month, 6-months, and 12-months). EEG also will be collected at the 1-month, 6-month, and 12-month assessments, and MRI will be collected at the 6-month and 12-month assessments.

ELIGIBILITY:
Inclusion Criteria:

* Veterans of Post-9/11 military conflicts
* with diagnosis of PTSD based on CAPS-5 related to Post-9/11 military combat

Exclusion Criteria:

* current enrollment in an acute experimental treatment for PTSD or trauma-focused psychotherapy treatment
* PTSD-inducing trauma exposure occurring within the last 3 months prior to pre-enrollment evaluation
* history of epilepsy or seizure disorder, a history of major head trauma,
* any neurologic condition likely to increase risk of seizures,
* brain tumors,
* moderate to severe substance use disorder in last 3 months or any substance use that puts the participant at increased risk or significant impairment
* stroke, and blood vessel abnormalities in the brain,
* dementia,
* Parkinson's disease, Huntington's chorea, or multiple sclerosis
* a high suicide risk
* a lifetime history of psychotic disorder or bipolar disorder
* inability to stop taking any medication that significantly lowers the seizure threshold
* pregnant or nursing
* metal fragments in the head, or any metal objects in or near the head that cannot be safely removed
* We will screen for a history of traumatic brain injury and exclude potential participants from the study if they have a history of severe TBI or are at high risk for seizures.
* history of seizures
* non-English speakers because not all of the screening forms, questionnaires, and tests are available in any language except for English
* cardiac pacemaker, implanted medication pumps of any sort that would increase the risk of rTMS
* any current medical condition that could preclude being able to safely participate in TMS treatment,
* use of prescription medication or illegal substances that lower the seizure threshold
* previous rTMS

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 330 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Treatment group differences in change from baseline to 6-months post-treatment on the Clinician Administered Posttraumatic Stress Disorder Scale for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (CAPS-5) Total Severity Score | Outcome measures will be measured twice over a period of 37 weeks: Baseline, 6-Month Post-Treatment
  Evaluation of treatment group differences on the Clinician Administered Posttraumatic Stress Disorder Scale for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (CAPS-5) Total Severity Score (20 item sum, range 0-80, higher score=greater severity) in change from baseline to 6 months after the 12-week interventions.
  Weathers, FW, Blake, DD, Schnurr, PP, Kaloupek, DG, Marx, BP, & Keane, TM. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). www.ptsd.va.gov: National Center for PTSD, 2013.

SECONDARY OUTCOMES:
Treatment group differences in change from baseline to 1 month post-treatment on the Clinician Administered Posttraumatic Stress Disorder Scale for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (CAPS-5) Total Severity Score | Outcome measures will be measured twice over a period of 17 weeks: Baseline, 1-Month Post-Treatment
  Evaluation of treatment group differences on the Clinician Administered Posttraumatic Stress Disorder Scale for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (CAPS-5) Total Severity Score (20 item sum, range 0-80, higher score=greater severity) in change from baseline to 1 month after the 12-week interventions.
  Weathers, FW, Blake, DD, Schnurr, PP, Kaloupek, DG, Marx, BP, & Keane, TM. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). www.ptsd.va.gov: National Center for PTSD, 2013.
Treatment group differences in change from baseline to 12 months post-treatment on the Clinician Administered Posttraumatic Stress Disorder Scale for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (CAPS-5) Total Severity Score | Outcome measures will be measured twice over a period of 61 weeks: Baseline, 12-Month Post-Treatment
  Evaluation of treatment group differences on the Clinician Administered Posttraumatic Stress Disorder Scale for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (CAPS-5) Total Severity Score (20 item sum, range 0-80, higher score=greater severity) in change from baseline to 12 months after the 12-week interventions.
  Weathers, FW, Blake, DD, Schnurr, PP, Kaloupek, DG, Marx, BP, & Keane, TM. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). www.ptsd.va.gov: National Center for PTSD, 2013.
Treatment group differences in change from baseline to 1 month post-treatment on the Posttraumatic Stress Disorder Checklist for for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (PCL-5) Total Severity Score | Outcome measures will be measured twice over a period of 17 weeks: Baseline, 1-Month Post-Treatment
  Evaluation of treatment group differences on the Posttraumatic Stress Disorder Checklist for for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (PCL-5) Total Severity Score (20 item sum, range 0-80, higher score=greater severity) in change from baseline to 1 month after the 12-week interventions.
  Weathers FW, Litz BT, Keane TM, Palmieri PA, Marx BP, Schnurr PP. The PTSD Checklist for DSM-5 (PCL-5). Scale available from the National Center for PTSD at www.ptsd.va.gov, 2013.
Treatment group differences in change from baseline to 6 months post-treatment on the Posttraumatic Stress Disorder Checklist for for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (PCL-5) Total Severity Score | Outcome measures will be measured twice over a period of 37 weeks: Baseline, 6-Month Post-Treatment
  Evaluation of treatment group differences on the Posttraumatic Stress Disorder Checklist for for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (PCL-5) Total Severity Score (20 item sum, range 0-80, higher score=greater severity) in change from baseline to 6 months after the 12-week interventions.
  Weathers FW, Litz BT, Keane TM, Palmieri PA, Marx BP, Schnurr PP. The PTSD Checklist for DSM-5 (PCL-5). Scale available from the National Center for PTSD at www.ptsd.va.gov, 2013.
Treatment group differences in change from baseline to 12 months post-treatment on the Posttraumatic Stress Disorder Checklist for for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (PCL-5) Total Severity Score | Outcome measures will be measured twice over a period of 61 weeks: Baseline, 12-Month Post-Treatment
  Evaluation of treatment group differences on the Posttraumatic Stress Disorder Checklist for for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (PCL-5) Total Severity Score (20 item sum, range 0-80, higher score=greater severity) in change from baseline to 12 months after the 12-week interventions.
  Weathers FW, Litz BT, Keane TM, Palmieri PA, Marx BP, Schnurr PP. The PTSD Checklist for DSM-5 (PCL-5). Scale available from the National Center for PTSD at www.ptsd.va.gov, 2013.
Treatment group differences in change from baseline to 1 month post-treatment on the Clinician Administered Posttraumatic Stress Disorder Scale for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (CAPS-5) Symptom Cluster Scores | Outcome measures will be measured twice over a period of 17 weeks: Baseline, 1-Month Post-Treatment
  Evaluation of treatment group differences on Clinician Administered Posttraumatic Stress Disorder Scale for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (CAPS-5) Symptom Cluster Scores (cluster item sum, higher scores=greater severity) in change from baseline to 1 month after the 12-week interventions. Evaluations of 4-Symptom Cluster Model ([1] Intrusions, range 0-20, [2] Avoidance, range 0-8, [3] Negative Cognition/Mood, range 0-28, and [4] Arousal/Reactivity, range 0-24) and 7-Symptom Cluster Model ([1] Intrusions, range 0-20, [2] Avoidance, range 0-8, [3] Negative Affect, range 0-16), [4] Anhedonia, range 0-12, [5] Externalizing, range 0-8, [6] Anxious Arousal, range 0-8, and [7] Dysphoric Arousal, range 0-8).
  Weathers FW, Bovin MJ, Lee DJ, Sloan DM, Schnurr PP, Kaloupek DG, Keane TM, Marx BP. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5): Development and initial psychometric evaluation in military veterans. Psychol Assess 30(3):383-395, 2018.
Treatment group differences in change from baseline to 6 months post-treatment on the Clinician Administered Posttraumatic Stress Disorder Scale for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (CAPS-5) Symptom Cluster Scores | Outcome measures will be measured twice over a period of 37 weeks: Baseline, 6-Month Post-Treatment
  Evaluation of treatment group differences on Clinician Administered Posttraumatic Stress Disorder Scale for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (CAPS-5) Symptom Cluster Scores (cluster item sum, higher scores=greater severity) in change from baseline to 6 months after the 12-week interventions. Evaluations of 4-Symptom Cluster Model ([1] Intrusions, range 0-20, [2] Avoidance, range 0-8, [3] Negative Cognition/Mood, range 0-28, and [4] Arousal/Reactivity, range 0-24) and 7-Symptom Cluster Model ([1] Intrusions, range 0-20, [2] Avoidance, range 0-8, [3] Negative Affect, range 0-16), [4] Anhedonia, range 0-12, [5] Externalizing, range 0-8, [6] Anxious Arousal, range 0-8, and [7] Dysphoric Arousal, range 0-8).
  Weathers FW, Bovin MJ, Lee DJ, Sloan DM, Schnurr PP, Kaloupek DG, Keane TM, Marx BP. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5): Development and initial psychometric evaluation in military veterans. Psychol Assess 30(3):383-395, 2018.
Treatment group differences in change from baseline to 12 months post-treatment on the Clinician Administered Posttraumatic Stress Disorder Scale for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (CAPS-5) Symptom Cluster Scores | Outcome measures will be measured twice over a period of 61 weeks: Baseline, 12-Month Post-Treatment
  Evaluation of treatment group differences on Clinician Administered Posttraumatic Stress Disorder Scale for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (CAPS-5) Symptom Cluster Scores (cluster item sum, higher scores=greater severity) in change from baseline to 12 months after the 12-week intervention. Evaluations of 4-Symptom Cluster Model ([1] Intrusions, range 0-20, [2] Avoidance, range 0-8, [3] Negative Cognition/Mood, range 0-28, and [4] Arousal/Reactivity, range 0-24) and 7-Symptom Cluster Model ([1] Intrusions, range 0-20, [2] Avoidance, range 0-8, [3] Negative Affect, range 0-16), [4] Anhedonia, range 0-12, [5] Externalizing, range 0-8, [6] Anxious Arousal, range 0-8, and [7] Dysphoric Arousal, range 0-8).
  Weathers FW, Bovin MJ, Lee DJ, Sloan DM, Schnurr PP, Kaloupek DG, Keane TM, Marx BP. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5): Development and initial psychometric evaluation in military veterans. Psychol Assess 30(3):383-395, 2018.
Treatment group differences in change from baseline to 6 weeks (5th intervention session) on the Clinician Administered Posttraumatic Stress Disorder Scale for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (CAPS-5) Total Score | Outcome measures will be measured twice over a period of 6 weeks: Baseline, 6 weeks
  Evaluation of treatment group differences on the Clinician Administered Posttraumatic Stress Disorder Scale for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (CAPS-5) Total Severity Score (20 item sum, range 0-80, higher score=greater severity) in change from baseline to 6 weeks.
  Weathers, F.W., Blake, D.D., Schnurr, P.P., Kaloupek, D.G., Marx, B.P., & Keane, T.M. (2013). The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). Interview available from the National Center for PTSD at www.ptsd.va.gov.
Treatment group differences in change from baseline to 10 weeks (9th intervention session) on the Clinician Administered Posttraumatic Stress Disorder Scale for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (CAPS-5) Total Score | Outcome measures will be measured twice over a period of 10 weeks: Baseline, 10 weeks
  Evaluation of treatment group differences on the Clinician Administered Posttraumatic Stress Disorder Scale for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (CAPS-5) Total Severity Score (20 item sum, range 0-80, higher score=greater severity) in change from baseline to 10 weeks.
  Weathers, F.W., Blake, D.D., Schnurr, P.P., Kaloupek, D.G., Marx, B.P., & Keane, T.M. (2013). The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). Interview available from the National Center for PTSD at www.ptsd.va.gov.
Treatment group differences in change from baseline to 6 weeks (5th intervention session) on the Clinician Administered Posttraumatic Stress Disorder Scale for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (CAPS-5) Symptom Cluster | Outcome measures will be measured twice over a period of 6 weeks: Baseline, 6 weeks
  Evaluation of treatment group differences on Clinician Administered Posttraumatic Stress Disorder Scale for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (CAPS-5) Symptom Cluster Scores (cluster item sum, higher scores=greater severity) in change from baseline to 6 weeks. Evaluations of 4-Symptom Cluster Model ([1] Intrusions, range 0-20, [2] Avoidance, range 0-8, [3] Negative Cognition/Mood, range 0-28, and [4] Arousal/Reactivity, range 0-24) and 7-Symptom Cluster Model ([1] Intrusions, range 0-20, [2] Avoidance, range 0-8, [3] Negative Affect, range 0-16), [4] Anhedonia, range 0-12, [5] Externalizing, range 0-8, [6] Anxious Arousal, range 0-8, and [7] Dysphoric Arousal, range 0-8).
  Weathers FW, Bovin MJ, Lee DJ, Sloan DM, Schnurr PP, Kaloupek DG, Keane TM, Marx BP. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5): Development and initial psychometric evaluation in military veterans. Psychol Assess 30(3):383-395, 2018.
Treatment group differences in change from baseline to 10 weeks (9th intervention session) on the Clinician Administered Posttraumatic Stress Disorder Scale for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (CAPS-5) Symptom Clust | Outcome measures will be measured twice over a period of 10 weeks: Baseline, 10 weeks
  Evaluation of treatment group differences on Clinician Administered Posttraumatic Stress Disorder Scale for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (CAPS-5) Symptom Cluster Scores (cluster item sum, higher scores=greater severity) in change from baseline to 10 weeks. Evaluations of 4-Symptom Cluster Model ([1] Intrusions, range 0-20, [2] Avoidance, range 0-8, [3] Negative Cognition/Mood, range 0-28, and [4] Arousal/Reactivity, range 0-24) and 7-Symptom Cluster Model ([1] Intrusions, range 0-20, [2] Avoidance, range 0-8, [3] Negative Affect, range 0-16), [4] Anhedonia, range 0-12, [5] Externalizing, range 0-8, [6] Anxious Arousal, range 0-8, and [7] Dysphoric Arousal, range 0-8).
  Weathers FW, Bovin MJ, Lee DJ, Sloan DM, Schnurr PP, Kaloupek DG, Keane TM, Marx BP. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5): Development and initial psychometric evaluation in military veterans. Psychol Assess 30(3):383-395, 2018.
Treatment group differences in change from baseline to 1 month post-treatment on the Posttraumatic Stress Disorder Checklist for for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (PCL-5) Symptom Cluster Scores | Outcome measures will be measured twice over a period of 17 weeks: Baseline, 1-Month Post-Treatment
  Evaluation of treatment group differences on Posttraumatic Stress Disorder Checklist for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (PCL-5) Symptom Cluster Scores (cluster item sum, higher scores=greater severity) in change from baseline to 1 month after 12-week interventions. Evaluations of 4-Symptom Cluster Model ([1] Intrusions, range 0-20, [2] Avoidance, range 0-8, [3] Negative Cognition/Mood, range 0-28, and [4] Arousal/Reactivity, range 0-24) and 7-Symptom Cluster Model ([1] Intrusions, range 0-20, [2] Avoidance, range 0-8, [3] Negative Affect, range 0-16), [4] Anhedonia, range 0-12, [5] Externalizing, range 0-8, [6] Anxious Arousal, range 0-8, and [7] Dysphoric Arousal, range 0-8).
  Bovin, MJ, Marx, BP, Weathers, FW, Gallagher, MW, Rodriguez, P, Schnurr, PP, Keane, TM. Psychometric properties of the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (PCL-5) in Veterans. Psychol Assess 28(11):1379-1391, 2016.
Treatment group differences in change from baseline to 6 months post-treatment on the Posttraumatic Stress Disorder Checklist for for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (PCL-5) Symptom Cluster Scores | Outcome measures will be measured twice over a period of 37 weeks: Baseline, 6-Month Post-Treatment
  Evaluation of treatment group differences on Posttraumatic Stress Disorder Checklist for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (PCL-5) Symptom Cluster Scores (cluster item sum, higher scores=greater severity) in change from baseline to 6 months after 12-week interventions. Evaluations of 4-Symptom Cluster Model ([1] Intrusions, range 0-20, [2] Avoidance, range 0-8, [3] Negative Cognition/Mood, range 0-28, and [4] Arousal/Reactivity, range 0-24) and 7-Symptom Cluster Model ([1] Intrusions, range 0-20, [2] Avoidance, range 0-8, [3] Negative Affect, range 0-16), [4] Anhedonia, range 0-12, [5] Externalizing, range 0-8, [6] Anxious Arousal, range 0-8, and [7] Dysphoric Arousal, range 0-8).
  Bovin, MJ, Marx, BP, Weathers, FW, Gallagher, MW, Rodriguez, P, Schnurr, PP, Keane, TM. Psychometric properties of the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (PCL-5) in Veterans. Psychol Assess 28(11):1379-1391, 2016.
Treatment group differences in change from baseline to 12 months post-treatment on the Posttraumatic Stress Disorder Checklist for for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (PCL-5) Symptom Cluster Scores | Outcome measures will be measured twice over a period of 61 weeks: Baseline, 12-Month Post-Treatment
  Evaluation of treatment group differences on Posttraumatic Stress Disorder Checklist for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (PCL-5) Symptom Cluster Scores (cluster item sum, higher scores=greater severity) in change from baseline to 12 months after 12-week interventions. Evaluations of 4-Symptom Cluster Model ([1] Intrusions, range 0-20, [2] Avoidance, range 0-8, [3] Negative Cognition/Mood, range 0-28, and [4] Arousal/Reactivity, range 0-24) and 7-Symptom Cluster Model ([1] Intrusions, range 0-20, [2] Avoidance, range 0-8, [3] Negative Affect, range 0-16), [4] Anhedonia, range 0-12, [5] Externalizing, range 0-8, [6] Anxious Arousal, range 0-8, and [7] Dysphoric Arousal, range 0-8).
  Bovin, MJ, Marx, BP, Weathers, FW, Gallagher, MW, Rodriguez, P, Schnurr, PP, Keane, TM. Psychometric properties of the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (PCL-5) in Veterans. Psychol Assess 28(11):1379-1391, 2016.
Treatment group differences in change from baseline to 6 weeks (5th intervention session) on the Posttraumatic Stress Disorder Checklist for for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (PCL-5) Symptom Cluster Scores | Outcome measures will be measured twice over a period of 6 weeks: Baseline, 6 weeks
  Evaluation of treatment group differences on Posttraumatic Stress Disorder Checklist for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (PCL-5) Symptom Cluster Scores (cluster item sum, higher scores=greater severity) in change from baseline to 6 weeks. Evaluations of 4-Symptom Cluster Model ([1] Intrusions, range 0-20, [2] Avoidance, range 0-8, [3] Negative Cognition/Mood, range 0-28, and [4] Arousal/Reactivity, range 0-24) and 7-Symptom Cluster Model ([1] Intrusions, range 0-20, [2] Avoidance, range 0-8, [3] Negative Affect, range 0-16), [4] Anhedonia, range 0-12, [5] Externalizing, range 0-8, [6] Anxious Arousal, range 0-8, and [7] Dysphoric Arousal, range 0-8).
  Bovin, MJ, Marx, BP, Weathers, FW, Gallagher, MW, Rodriguez, P, Schnurr, PP, Keane, TM. Psychometric properties of the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (PCL-5) in Veterans. Psychol Assess 28(11):1379-1391, 2016.
Treatment group differences in change from baseline to 10 weeks (9th intervention session) on the Posttraumatic Stress Disorder Checklist for for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (PCL-5) Symptom Cluster Scores | Outcome measures will be measured twice over a period of 10 weeks: Baseline, 10 weeks
  Evaluation of treatment group differences on Posttraumatic Stress Disorder Checklist for Diagnostic and Statistical Manual of Mental Disorders (5th edition) (PCL-5) Symptom Cluster Scores (cluster item sum, higher scores=greater severity) in change from baseline to 10 weeks. Evaluations of 4-Symptom Cluster Model ([1] Intrusions, range 0-20, [2] Avoidance, range 0-8, [3] Negative Cognition/Mood, range 0-28, and [4] Arousal/Reactivity, range 0-24) and 7-Symptom Cluster Model ([1] Intrusions, range 0-20, [2] Avoidance, range 0-8, [3] Negative Affect, range 0-16), [4] Anhedonia, range 0-12, [5] Externalizing, range 0-8, [6] Anxious Arousal, range 0-8, and [7] Dysphoric Arousal, range 0-8).
  Bovin, MJ, Marx, BP, Weathers, FW, Gallagher, MW, Rodriguez, P, Schnurr, PP, Keane, TM. Psychometric properties of the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (PCL-5) in Veterans. Psychol Assess 28(11):1379-1391, 2016.
Treatment group differences in change from baseline to 1 month post-treatment on the Mississippi Scale for Combat Related Posttraumatic Stress Disorder | Outcome measures will be measured twice over a period of 17 weeks: Baseline, 1-Month Post-Treatment
  Evaluation of treatment group differences on the Mississippi Scale for Combat Related Posttraumatic Stress Disorder Total Score (35 item sum, range 35-175, higher score=greater severity) in change from baseline to 1-month after the 12-week interventions.
  Keane TM, Caddell JM, Taylor KL. Mississippi Scale for Combat-Related Posttraumatic Stress Disorder: three studies in reliability and validity. J Consult Clin Psychol 56(1):85-90, 1988.
Treatment group differences in change from baseline to 6 months post-treatment on the Mississippi Scale for Combat Related Posttraumatic Stress Disorder | Outcome measures will be measured twice over a period of 37 weeks: Baseline, 6-Month Post-Treatment
  Evaluation of treatment group differences on the Mississippi Scale for Combat Related Posttraumatic Stress Disorder Total Score (35 item sum, range 35-175, higher score=greater severity) in change from baseline to 6-months after the 12-week interventions.
  Keane TM, Caddell JM, Taylor KL. Mississippi Scale for Combat-Related Posttraumatic Stress Disorder: three studies in reliability and validity. J Consult Clin Psychol 56(1):85-90, 1988.
Treatment group differences in change from baseline to 12 months post-treatment on the Mississippi Scale for Combat Related Posttraumatic Stress Disorder | Outcome measures will be measured twice over a period of 61 weeks: Baseline, 12-Month Post-Treatment
  Evaluation of treatment group differences on the Mississippi Scale for Combat Related Posttraumatic Stress Disorder Total Score (35 item sum, range 35-175, higher score=greater severity) in change from baseline to 12-months after the 12-week interventions.
  Keane TM, Caddell JM, Taylor KL. Mississippi Scale for Combat-Related Posttraumatic Stress Disorder: three studies in reliability and validity. J Consult Clin Psychol 56(1):85-90, 1988.
Treatment group differences in change from baseline to 1 month post-treatment on Montgomery Asberg Depression Rating Scale | Outcome measures will be measured twice over a period of 17 weeks: Baseline, 1-Month Post-Treatment
  Evaluation of treatment group differences on the Montgomery Asberg Depression Rating Scale (10 item sum, range 0-60, higher score=greater severity) in change from baseline to 1-month after the 12-week interventions.
  Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry 134:382-389, 1979.
Treatment group differences in change from baseline to 6 months post-treatment on Montgomery Asberg Depression Rating Scale | Outcome measures will be measured twice over a period of 37 weeks: Baseline, 6-Month Post-Treatment
  Evaluation of treatment group differences on the Montgomery Asberg Depression Rating Scale (10 item sum, range 0-60, higher score=greater severity) in change from baseline to 6-months after the 12-week interventions.
  Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry 134:382-389, 1979.
Treatment group differences in change from baseline to 12 months post-treatment on Montgomery Asberg Depression Rating Scale | Outcome measures will be measured twice over a period of 61 weeks: Baseline, 12-Month Post-Treatment
  Evaluation of treatment group differences on the Montgomery Asberg Depression Rating Scale (10 item sum, range 0-60, higher score=greater severity) in change from baseline to 12-months after the 12-week interventions.
  Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry 134:382-389, 1979.
Treatment group differences in change from baseline to 6 weeks (5th intervention session) on Montgomery Asberg Depression Rating Scale | Outcome measures will be measured twice over a period of 6 weeks: Baseline, 6 weeks
  Evaluation of treatment group differences on the Montgomery Asberg Depression Rating Scale (10 item sum, range 0-60, higher score=greater severity) in change from baseline to 6 weeks.
  Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry 134:382-389, 1979.
Treatment group differences in change from baseline to 10 weeks (9th intervention session) on Montgomery Asberg Depression Rating Scale | Outcome measures will be measured twice over a period of 10 weeks: Baseline, 10 weeks
  Evaluation of treatment group differences on the Montgomery Asberg Depression Rating Scale (10 item sum, range 0-60, higher score=greater severity) in change from baseline to 10 weeks.
  Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry 134:382-389, 1979.
Treatment group differences in change from baseline to 1 month post-treatment on the Quick Inventory of Depressive Symptomatology | Outcome measures will be measured twice over a period of 17 weeks: Baseline, 1-Month Post-Treatment
  Evaluation of treatment group differences on the Quick Inventory of Depressive Symptomatology (QIDS) (9 domain sum, range 0-27, higher score=greater severity) in change from baseline to 1-month after the 12-week interventions.
  Rush, AJ, Trivedi, MH, et al. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry 54(5):573-583, 2003.
Treatment group differences in change from baseline to 6 months post-treatment on the Quick Inventory of Depressive Symptomatology | Outcome measures will be measured twice over a period of 37 weeks: Baseline, 6-Month Post-Treatment
  Evaluation of treatment group differences on the Quick Inventory of Depressive Symptomatology (QIDS) (9 domain sum, range 0-27, higher score=greater severity) in change from baseline to 6-months after the 12-week interventions.
  Rush, AJ, Trivedi, MH, et al. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry 54(5):573-583, 2003.
Treatment group differences in change from baseline to 12 months post-treatment on the Quick Inventory of Depressive Symptomatology | Outcome measures will be measured twice over a period of 61 weeks: Baseline, 12-Month Post-Treatment
  Evaluation of treatment group differences on the Quick Inventory of Depressive Symptomatology (QIDS) (9 domain sum, range 0-27, higher score=greater severity) in change from baseline to 12-months after the 12-week interventions.
  Rush, AJ, Trivedi, MH, et al. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry 54(5):573-583, 2003.
Treatment group differences in change from baseline to 6 weeks (5th intervention session ) on the Quick Inventory of Depressive Symptomatology | Outcome measures will be measured twice over a period of 6 weeks: Baseline, 6 weeks
  Evaluation of treatment group differences on the Quick Inventory of Depressive Symptomatology (QIDS) (9 domain sum, range 0-27, higher score=greater severity) in change from baseline to 6 weeks.
  Rush, AJ, Trivedi, MH, et al. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry 54(5):573-583, 2003.
Treatment group differences from baseline to 10 weeks (9th intervention session) on the Quick Inventory of Depressive Symptomatology | Outcome measures will be measured twice over a period of 10 weeks: Baseline, 10 weeks
  Evaluation of treatment group differences on the Quick Inventory of Depressive Symptomatology (QIDS) (9 domain sum, range 0-27, higher score=greater severity) in change from baseline to 10 weeks.
  Rush, AJ, Trivedi, MH, et al. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry 54(5):573-583, 2003.
Treatment group differences in change from baseline to 1 month post-treatment on the Inventory of Psychosocial Functioning | Outcome measures will be measured twice over a period of 17 weeks: Baseline, 1-Month Post-Treatment
  Evaluation of treatment group differences on the Inventory of Psychosocial Functioning (IPF) Overall Score (mean of completed domain scores, range 0-100, higher score=greater impairment) in change from baseline to 1 month following the 12-week interventions.
  Bovin MJ, Black SK, Rodriguez P, Lunney CA, Kleiman SE, Weathers FW, Schnurr PP, Spira J, Keane TM, Marx BP. Development and validation of a measure of PTSD-related psychosocial functional impairment: The Inventory of Psychosocial Functioning. Psychol Serv 15(2):216-229, 2018.
Treatment group differences in change from baseline to 6 months post-treatment on the Inventory of Psychosocial Functioning | Outcome measures will be measured twice over a period of 37 weeks: Baseline, 6-Month Post-Treatment
  Evaluation of treatment group differences on the Inventory of Psychosocial Functioning (IPF) Overall Score (mean of completed domain scores, range 0-100, higher score=greater impairment) in change from baseline to 6 months after the 12-week interventions.
  Bovin MJ, Black SK, Rodriguez P, Lunney CA, Kleiman SE, Weathers FW, Schnurr PP, Spira J, Keane TM, Marx BP. Development and validation of a measure of PTSD-related psychosocial functional impairment: The Inventory of Psychosocial Functioning. Psychol Serv 15(2):216-229, 2018.
Treatment group differences in change from baseline to 12 months post-treatment on the Inventory of Psychosocial Functioning | Outcome measures will be measured twice over a period of 61 weeks: Baseline, 12-Month Post-Treatment
  Evaluation of treatment group differences on the Inventory of Psychosocial Functioning (IPF) Overall Score (mean of completed domain scores, range 0-100, higher score=greater impairment) in change from baseline to 12 months after the 12-week interventions.
  Bovin MJ, Black SK, Rodriguez P, Lunney CA, Kleiman SE, Weathers FW, Schnurr PP, Spira J, Keane TM, Marx BP. Development and validation of a measure of PTSD-related psychosocial functional impairment: The Inventory of Psychosocial Functioning. Psychol Serv 15(2):216-229, 2018.
Treatment group differences in change from baseline to 1 month post-treatment on the Short Impulsive Behavior Scale | Outcome measures will be measured twice over a period of 17 weeks: Baseline, 1-Month Post-Treatment
  Evaluation of treatment group differences on the Short Impulsive Behavior Scale (UPPS-P) Total Score (mean item rating, range 1-4, higher score=greater impulsivity) in change from baseline to 1 month after the 12-week interventions.
  Cyders MA, Littlefield AK, Coffey S, Karyadi KA. Examination of a short English version of the UPPS-P Impulsive Behavior Scale. Addict Behav 39(9):1372-1376, 2014.
Treatment group differences in change from baseline to 6 months post-treatment on the Short Impulsive Behavior Scale | Outcome measures will be measured twice over a period of 37 weeks: Baseline, 6-Month Post-Treatment
  Evaluation of treatment group differences on the Short Impulsive Behavior Scale (UPPS-P) Total Score (mean item rating, range 1-4, higher score=greater impulsivity) in change from baseline to 6 months after the 12-week interventions.
  Cyders MA, Littlefield AK, Coffey S, Karyadi KA. Examination of a short English version of the UPPS-P Impulsive Behavior Scale. Addict Behav 39(9):1372-1376, 2014.
Treatment group differences in change from baseline to 12 months post-treatment on the Short Impulsive Behavior Scale | Outcome measures will be measured twice over a period of 61 weeks: Baseline, 12-Month Post-Treatment
  Evaluation of treatment group differences on the Short Impulsive Behavior Scale (UPPS-P) Total Score (mean item rating, range 1-4, higher score=greater impulsivity) in change from baseline to 12 months after the 12-week interventions.
  Cyders MA, Littlefield AK, Coffey S, Karyadi KA. Examination of a short English version of the UPPS-P Impulsive Behavior Scale. Addict Behav 39(9):1372-1376, 2014.
Treatment group differences in change from baseline to 1 month post-treatment on the Short Impulsive Behavior Subscales | Outcome measures will be measured twice over a period of 17 weeks: Baseline, 1-Month Post-Treatment
  Evaluation of treatment group differences on the Short Impulsive Behavior Scale (UPPS-P) Subscale Scores (mean item rating, range 1-4, higher score=greater impulsivity) in change from baseline to 1 month after the 12-week interventions. Evaluations on (1) Negative Urgency, (2) Perseverance, (3) Premeditation, (4) Sensation Seeking, and (5) Positive Urgency
  Cyders MA, Littlefield AK, Coffey S, Karyadi KA. Examination of a short English version of the UPPS-P Impulsive Behavior Scale. Addict Behav 39(9):1372-1376, 2014.
Treatment group differences in change from baseline to 6 months post-treatment on the Short Impulsive Behavior Subscales | Outcome measures will be measured twice over a period of 37 weeks: Baseline, 6-Month Post-Treatment
  Evaluation of treatment group differences on the Short Impulsive Behavior Scale (UPPS-P) Subscale Scores (mean item rating, range 1-4, higher score=greater impulsivity) in change from baseline to 6 months after the 12-week interventions. Evaluations on (1) Negative Urgency, (2) Perseverance, (3) Premeditation, (4) Sensation Seeking, and (5) Positive Urgency
  Cyders MA, Littlefield AK, Coffey S, Karyadi KA. Examination of a short English version of the UPPS-P Impulsive Behavior Scale. Addict Behav 39(9):1372-1376, 2014.
Treatment group differences in change from baseline to 12 months post-treatment on the Short Impulsive Behavior Subscales | Outcome measures will be measured twice over a period of 61 weeks: Baseline, 12-Month Post-Treatment
  Evaluation of treatment group differences on the Short Impulsive Behavior Scale (UPPS-P) Subscale Scores (mean item rating, range 1-4, higher score=greater impulsivity) in change from baseline to 12 months after the 12-week interventions. Evaluations on (1) Negative Urgency, (2) Perseverance, (3) Premeditation, (4) Sensation Seeking, and (5) Positive Urgency
  Cyders MA, Littlefield AK, Coffey S, Karyadi KA. Examination of a short English version of the UPPS-P Impulsive Behavior Scale. Addict Behav 39(9):1372-1376, 2014.
Treatment group differences in change in aggression from baseline to 1 month post-treatment on the Buss-Perry Aggression Questionnaire | Outcome measures will be measured twice over a period of 17 weeks: Baseline, 1-Month Post-Treatment
  Evaluation of treatment group differences on the Buss-Perry Aggression Questionnaire Total Score (29 item sum, range 29-145, higher score=greater aggression) in change from baseline to 1 month after the 12-week interventions.
  Buss AH, Perry M. The Aggression Questionnaire. J Pers Soc Psychol 63(3):452-459, 1992.
Treatment group differences in change from baseline to 6 months post-treatment on the Buss-Perry Aggression Questionnaire | Outcome measures will be measured twice over a period of 37 weeks: Baseline, 6-Month Post-Treatment
  Evaluation of treatment group differences on the Buss-Perry Aggression Questionnaire Total Score (29 item sum, range 29-145, higher score=greater aggression) in change from baseline to 6 months after the 12-week interventions.
  Buss AH, Perry M. The Aggression Questionnaire. J Pers Soc Psychol 63(3):452-459, 1992.
Treatment group differences in change from baseline to 12 months post-treatment on the Buss-Perry Aggression Questionnaire | Outcome measures will be measured twice over a period of 61 weeks: Baseline, 12-Month Post-Treatment
  Evaluation of treatment group differences on the Buss-Perry Aggression Questionnaire Total Score (29 item sum, range 29-145, higher score=greater aggression) in change from baseline to 12 months after the 12-week interventions.
  Buss AH, Perry M. The Aggression Questionnaire. J Pers Soc Psychol 63(3):452-459, 1992.
Treatment group differences in change from baseline to 1 month post-treatment on the Buss-Perry Aggression Questionnaire Subscales | Outcome measures will be measured twice over a period of 17 weeks: Baseline, 1-Month Post-Treatment
  Evaluation of treatment group differences on the Buss-Perry Aggression Questionnaire Subscale Scores (subscale item sum, higher score=greater aggression) in change from baseline to 1 month after the 12-week interventions. Evaluated on: Physical Aggression (9 items, range 9-45), Verbal Aggression (5 items, range 5-25), Anger (7 items, range 7-35), and Hostility (8 items, range 8-40).
  Buss AH, Perry M. The Aggression Questionnaire. J Pers Soc Psychol 63(3):452-459, 1992.
Treatment group differences in change from baseline to 6 months post-treatment on the Buss-Perry Aggression Questionnaire Subscales | Outcome measures will be measured twice over a period of 37 weeks: Baseline, 6-Month Post-Treatment
  Evaluation of treatment group differences on the Buss-Perry Aggression Questionnaire Subscale Scores (subscale item sum, higher score=greater aggression) in change from baseline to 6 months after the 12-week interventions. Evaluated on: Physical Aggression (9 items, range 9-45), Verbal Aggression (5 items, range 5-25), Anger (7 items, range 7-35), and Hostility (8 items, range 8-40).
  Buss AH, Perry M. The Aggression Questionnaire. J Pers Soc Psychol 63(3):452-459, 1992.
Treatment group differences in change from baseline to 12 months post-treatment on the Buss-Perry Aggression Questionnaire Subscales | Outcome measures will be measured twice over a period of 61 weeks: Baseline, 12-Month Post-Treatment
  Evaluation of treatment group differences on the Buss-Perry Aggression Questionnaire Subscale Scores (subscale item sum, higher score=greater aggression) in change from baseline to 12 months after the 12-week interventions. Evaluated on: Physical Aggression (9 items, range 9-45), Verbal Aggression (5 items, range 5-25), Anger (7 items, range 7-35), and Hostility (8 items, range 8-40).
  Buss AH, Perry M. The Aggression Questionnaire. J Pers Soc Psychol 63(3):452-459, 1992.
Treatment group differences in change from baseline to 1 month post-treatment in event-related potential in response to trauma-specific auditory stimuli | Outcome measures will be measured twice over a period of 17 weeks: Baseline, 1-Month Post-Treatment
  Evaluation of treatment group differences in change from baseline to 1 month following the 12-week interventions in event-related potential (ERP) on trauma-specific threatening auditory stimuli compared to non-specific threatening and non-threatening auditory stimuli. Measured as change in microvolts separately on the N2 and P3 ERP components.
  Tillman GD et al. Repetitive transcranial magnetic stimulation and threat memory: selective reduction of combat threat memory p300 response after right frontal-lobe stimulation. J Neuropsychiatry Clin Neurosci 23(1):40-7, 2011.
Treatment group differences in change from baseline to 6 months post-treatment in event-related potential in response to trauma-specific auditory stimuli | Outcome measures will be measured twice over a period of 37 weeks: Baseline, 6-Month Post-Treatment
  Evaluation of treatment group differences in change from baseline to 6 months following the 12-week interventions in event-related potential (ERP) on trauma-specific threatening auditory stimuli compared to non-specific threatening and non-threatening auditory stimuli. Measured as change in microvolts separately on the N2 and P3 ERP components.
  Tillman GD et al. Repetitive transcranial magnetic stimulation and threat memory: selective reduction of combat threat memory p300 response after right frontal-lobe stimulation. J Neuropsychiatry Clin Neurosci 23(1):40-7, 2011.
Treatment group differences in change from baseline to 12 months post-treatment in event-related potential in response to trauma-specific auditory stimuli | Outcome measures will be measured twice over a period of 61 weeks: Baseline, 12-Month Post-Treatment
  Evaluation of treatment group differences in change from baseline to 12 months following the 12-week interventions in event-related potential (ERP) on trauma-specific threatening auditory stimuli compared to non-specific threatening and non-threatening auditory stimuli. Measured as change in microvolts separately on the N2 and P3 ERP components.
  Tillman GD et al. Repetitive transcranial magnetic stimulation and threat memory: selective reduction of combat threat memory p300 response after right frontal-lobe stimulation. J Neuropsychiatry Clin Neurosci 23(1):40-7, 2011.
Treatment group differences in change from baseline to 1 month post-treatment in event-related potential in response to trauma-specific visual stimuli | Outcome measures will be measured twice over a period of 17 weeks: Baseline, 1-Month Post-Treatment
  Evaluation of treatment group differences in change from baseline to 1 month following the 12-week interventions in event-related potential (ERP) on trauma-specific visual stimuli compared to non-specific threatening and non-threatening visual stimuli. Measured as change in microvolts separately on the N2 and P3 ERP components.
  DeLaRosa BL et al. Electrophysiological spatiotemporal dynamics during implicit visual threat processing. Brain Cogn 91:54-61, 2014.
Treatment group differences in change from baseline to 6 months post-treatment in event-related potential in response to trauma-specific visual stimuli | Outcome measures will be measured twice over a period of 37 weeks: Baseline, 6-Month Post-Treatment
  Evaluation of treatment group differences in change from baseline to 6 months following the 12-week interventions in event-related potential (ERP) on trauma-specific visual stimuli compared to non-specific threatening and non-threatening visual stimuli. Measured as change in microvolts separately on the N2 and P3 ERP components.
  DeLaRosa BL et al. Electrophysiological spatiotemporal dynamics during implicit visual threat processing. Brain Cogn 91:54-61, 2014.
Treatment group differences in change from baseline to 12 months post-treatment in event-related potential in response to trauma-specific visual stimuli | Outcome measures will be measured twice over a period of 61 weeks: Baseline, 12-Month Post-Treatment
  Evaluation of treatment group differences in change from baseline to 12 months following the 12-week interventions in event-related potential (ERP) on trauma-specific visual stimuli compared to non-specific threatening and non-threatening visual stimuli. Measured as change in microvolts separately on the N2 and P3 ERP components.
  DeLaRosa BL et al. Electrophysiological spatiotemporal dynamics during implicit visual threat processing. Brain Cogn 91:54-61, 2014.
Treatment group differences in change from baseline to 1 month post-treatment in electroencephalography power in response to trauma-specific auditory stimuli | Outcome measures will be measured twice over a period of 17 weeks: Baseline, 1-Month Post-Treatment
  Evaluation of treatment group differences in change from baseline to 1 month following the 12-week interventions in change in electroencephalography (EEG) power within alpha- and theta-bands to trauma-specific threatening auditory stimuli compared to non-specific threatening and non-threatening auditory stimuli. For task conditions of interest, EEG power will be calculated separately at each electrode as log transformed, absolute power averages in the delta (1.5-3.5 Hz), theta (4-7.5 Hz), alpha (8-13 Hz), and beta (13.5-25 Hz) bands over time.
  Tillman GD et al. Repetitive transcranial magnetic stimulation and threat memory: selective reduction of combat threat memory p300 response after right frontal-lobe stimulation. J Neuropsychiatry Clin Neurosci 23(1):40-7, 2011.
Treatment group differences in change from baseline to 6 months post-treatment in electroencephalography power in response to trauma-specific auditory stimuli | Outcome measures will be measured twice over a period of 37 weeks: Baseline, 6-Month Post-Treatment
  Evaluation of treatment group differences in change from baseline to 6 months following the 12-week interventions in change in electroencephalography (EEG) power within alpha- and theta-bands to trauma-specific threatening auditory stimuli compared to non-specific threatening and non-threatening auditory stimuli. For task conditions of interest, EEG power will be calculated separately at each electrode as log transformed, absolute power averages in the delta (1.5-3.5 Hz), theta (4-7.5 Hz), alpha (8-13 Hz), and beta (13.5-25 Hz) bands over time.
  Tillman GD et al. Repetitive transcranial magnetic stimulation and threat memory: selective reduction of combat threat memory p300 response after right frontal-lobe stimulation. J Neuropsychiatry Clin Neurosci 23(1):40-7, 2011.
Treatment group differences in change from baseline to 12 months post-treatment in electroencephalography power in response to trauma-specific auditory stimuli | Outcome measures will be measured twice over a period of 61 weeks: Baseline, 12-Month Post-Treatment
  Evaluation of treatment group differences in change from baseline to 12 months following the 12-week interventions in change in electroencephalography (EEG) power within alpha- and theta-bands to trauma-specific threatening auditory stimuli compared to non-specific threatening and non-threatening auditory stimuli. For task conditions of interest, EEG power will be calculated separately at each electrode as log transformed, absolute power averages in the delta (1.5-3.5 Hz), theta (4-7.5 Hz), alpha (8-13 Hz), and beta (13.5-25 Hz) bands over time.
  Tillman GD et al. Repetitive transcranial magnetic stimulation and threat memory: selective reduction of combat threat memory p300 response after right frontal-lobe stimulation. J Neuropsychiatry Clin Neurosci 23(1):40-7, 2011.
Treatment group differences in change from baseline to 1 month post-treatment in electroencephalography power in response to trauma-specific visual stimuli | Outcome measures will be measured twice over a period of 17 weeks: Baseline, 1-Month Post-Treatment
  Evaluation of treatment group differences in change from baseline to 1 month following the 12-week interventions in change in electroencephalography (EEG) power within alpha- and theta-bands to trauma-specific visual stimuli compared to non-specific threatening and non-threatening visual stimuli. For task conditions of interest, EEG power will be calculated separately at each electrode as log transformed, absolute power averages in the delta (1.5-3.5 Hz), theta (4-7.5 Hz), alpha (8-13 Hz), and beta (13.5-25 Hz) bands over time.
  DeLaRosa BL et al. Electrophysiological spatiotemporal dynamics during implicit visual threat processing. Brain Cogn 91:54-61, 2014.
Treatment group differences in change from baseline to 6 months post-treatment in electroencephalography power in response to trauma-specific visual stimuli | Outcome measures will be measured twice over a period of 37 weeks: Baseline, 6-Month Post-Treatment
  Evaluation of treatment group differences in change from baseline to 6 months following the 12-week interventions in change in electroencephalography (EEG) power within alpha- and theta-bands to trauma-specific visual stimuli compared to non-specific threatening and non-threatening visual stimuli. For task conditions of interest, EEG power will be calculated separately at each electrode as log transformed, absolute power averages in the delta (1.5-3.5 Hz), theta (4-7.5 Hz), alpha (8-13 Hz), and beta (13.5-25 Hz) bands over time.
  DeLaRosa BL et al. Electrophysiological spatiotemporal dynamics during implicit visual threat processing. Brain Cogn 91:54-61, 2014.
Treatment group differences in change from baseline to 12 months post-treatment in electroencephalography power in response to trauma-specific visual stimuli | Outcome measures will be measured twice over a period of 61 weeks: Baseline, 12-Month Post-Treatment
  Evaluation of treatment group differences in change from baseline to 12 months following the 12-week interventions in change in electroencephalography (EEG) power within alpha- and theta-bands to trauma-specific visual stimuli compared to non-specific threatening and non-threatening visual stimuli. For task conditions of interest, EEG power will be calculated separately at each electrode as log transformed, absolute power averages in the delta (1.5-3.5 Hz), theta (4-7.5 Hz), alpha (8-13 Hz), and beta (13.5-25 Hz) bands over time.
  DeLaRosa BL et al. Electrophysiological spatiotemporal dynamics during implicit visual threat processing. Brain Cogn 91:54-61, 2014.
Treatment group differences in change from baseline to 1 month post-treatment in event-related potential responses in inhibitory control | Outcome measures will be measured twice over a period of 17 weeks: Baseline, 1-Month Post-Treatment
  Evaluation of treatment group differences in change from baseline to 1 month following the 12-week interventions in change in event-related potential (ERP) on inhibitory control trials (i.e., No-Go trials on the semantically cued inhibitory control task). Measured as change in microvolts separately on the N2 and P3 ERP components.
  Maguire MJ et al. The influence of perceptual and semantic categorization on inhibitory processing as measured by the N2-P3 response. Brain Cog 71; 196-203, 2009.
Treatment group differences in change from baseline to 6 months post-treatment in event-related potential responses in inhibitory control | Outcome measures will be measured twice over a period of 37 weeks: Baseline, 6-Month Post-Treatment
  Evaluation of treatment group differences in change from baseline to 6 months following the 12-week interventions in change in event-related potential (ERP) on inhibitory control trials (i.e., No-Go trials on the semantically cued inhibitory control task). Measured as change in microvolts separately on the N2 and P3 ERP components.
  Maguire MJ et al. The influence of perceptual and semantic categorization on inhibitory processing as measured by the N2-P3 response. Brain Cog 71; 196-203, 2009.
Treatment group differences in change from baseline to 12-month post-treatment in event-related potential responses in inhibitory control | Outcome measures will be measured twice over a period of 61 weeks: Baseline, 12-Month Post-Treatment
  Evaluation of treatment group differences in change from baseline to 12 months following the 12-week interventions in change in event-related potential (ERP) on inhibitory control trials (i.e., No-Go trials on the semantically cued inhibitory control task). Measured as change in microvolts separately on the N2 and P3 ERP components.
  Maguire MJ et al. The influence of perceptual and semantic categorization on inhibitory processing as measured by the N2-P3 response. Brain Cog 71; 196-203, 2009.
Treatment group differences in change from baseline to 1-month post-treatment in resting-state electroencephalography power | Outcome measures will be measured twice over a period of 17 weeks: Baseline, 1-Month Post-Treatment
  Evaluation of treatment group differences in change from baseline to 1 month following the 12-week interventions in change in resting-state electroencephalography (EEG) power. EEG power will be calculated separately at each electrode as the log transformed, absolute power in the delta (1.5-3.5 Hz), theta (4-7.5 Hz), alpha (8-13 Hz), and beta (13.5-25 Hz) bands for each eyes-open and eyes-closed epoch, and groups differences from baseline to 1-month in the average differences in the log transformed, absolute power between the eyes-open and eyes-closed conditions will be evaluated.
Treatment group differences in change from baseline to 6-months post-treatment in resting-state electroencephalography power | Outcome measures will be measured twice over a period of 37 weeks: Baseline, 6-Month Post-Treatment
  Evaluation of treatment group differences in change from baseline to 6 months following the 12-week interventions in change in resting-state electroencephalography (EEG) power. EEG power will be calculated separately at each electrode as the log transformed, absolute power in the delta (1.5-3.5 Hz), theta (4-7.5 Hz), alpha (8-13 Hz), and beta (13.5-25 Hz) bands for each eyes-open and eyes-closed epoch, and groups differences from baseline to 1-month in the average differences in the log transformed, absolute power between the eyes-open and eyes-closed conditions will be evaluated.
Treatment group differences in change from baseline to 12-months post-treatment in resting-state electroencephalography power | Outcome measures will be measured twice over a period of 61 weeks: Baseline, 12-Month Post-Treatment
  Evaluation of treatment group differences in change from baseline to 12 months following the 12-week interventions in change in resting-state electroencephalography (EEG) power. EEG power will be calculated separately at each electrode as the log transformed, absolute power in the delta (1.5-3.5 Hz), theta (4-7.5 Hz), alpha (8-13 Hz), and beta (13.5-25 Hz) bands for each eyes-open and eyes-closed epoch, and groups differences from baseline to 1-month in the average differences in the log transformed, absolute power between the eyes-open and eyes-closed conditions will be evaluated.
Treatment group differences in change from baseline to 6-months post-treatment trauma-specific responses in blood oxygen level dependent functional magnetic resonance imaging | Outcome measures will be measured twice over a period of 37 weeks: Baseline, 6-Month Post-Treatment
  Evaluation of treatment group differences from baseline to 6 months following the 12-week interventions in functional magnetic resonance imaging (fMRI) blood oxygen level dependent (BOLD) signal change (mean percent signal-change from the task baseline) to trauma-specific visual stimuli compared to non-specific threatening and non-threatening visual stimuli.
  Calley CS, et al. Threat as a feature in visual semantic object memory. Hum Brain Mapp. 34(8):1946-55, 2013.
Treatment group differences in change from baseline to 12 months post-treatment trauma-specific responses in blood oxygen level dependent functional magnetic resonance imaging | Outcome measures will be measured twice over a period of 61 weeks: Baseline, 12-Month Post-Treatment
  Evaluation of treatment group differences from baseline to 12 months following the 12-week interventions in functional magnetic resonance imaging (fMRI) blood oxygen level dependent (BOLD) signal change (mean percent signal-change from the task baseline) to trauma-specific visual stimuli compared to non-specific threatening and non-threatening visual stimuli.
  Calley CS, et al. Threat as a feature in visual semantic object memory. Hum Brain Mapp. 34(8):1946-55, 2013.
Treatment group differences in change from baseline to 6 months post-treatment in resting-state functional connectivity | Outcome measures will be measured twice over a period of 37 weeks: Baseline, 6-Month Post-Treatment
  Evaluation of treatment group differences from baseline to 6 months following the 12-week interventions in functional magnetic resonance imaging (fMRI) blood oxygen level dependent (BOLD) resting-state connectivity. Group differences in seed-based connectivity indices (mean standardized coherence parameter estimates) with right dorsolateral prefrontal cortex, amygdalae, thalamus, and dorsal anterior cingulate as the primary therapeutic targets will be calculated.
Treatment group differences in change from baseline to 12 months post-treatment in resting-state functional connectivity | Outcome measures will be measured twice over a period of 61 weeks: Baseline, 12-Month Post-Treatment
  Evaluation of treatment group differences from baseline to 12 months following the 12-week interventions in functional magnetic resonance imaging (fMRI) blood oxygen level dependent (BOLD) resting-state connectivity. Group differences in seed-based connectivity indices (mean standardized coherence parameter estimates) with right dorsolateral prefrontal cortex, amygdalae, thalamus, and dorsal anterior cingulate as the primary therapeutic targets will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: John Hart, Jr., MD, Principal Investigator — The University of Texas at Dallas; F. Andrew Kozel, MD, Principal Investigator — Florida State University, College of Medicine; John Burruss, MD, Principal Investigator — Metrocare Services of Dallas
Locations (3):
- United States (3):
  - Florida State University College of Medicine, Tallahassee, Florida
  - Metrocare Services of Dallas, Addison, Texas
  - The University of Texas at Dallas, Dallas, Texas

REFERENCES:
- [Background] Weathers FW, Bovin MJ, Lee DJ, Sloan DM, Schnurr PP, Kaloupek DG, Keane TM, Marx BP. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5): Development and initial psychometric evaluation in military veterans. Psychol Assess. 2018 Mar;30(3):383-395. doi: 10.1037/pas0000486. Epub 2017 May 11. PMID 28493729
- [Background] Weathers FW, Litz BT, Keane TM, Palmieri PA, Marx BP, Schnurr PP. The PTSD Checklist for DSM-5 (PCL-5). Scale available from the National Center for PTSD at www.ptsd.va.gov, 2013.
- [Background] Rush AJ, Trivedi MH, Ibrahim HM, Carmody TJ, Arnow B, Klein DN, Markowitz JC, Ninan PT, Kornstein S, Manber R, Thase ME, Kocsis JH, Keller MB. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry. 2003 Sep 1;54(5):573-83. doi: 10.1016/s0006-3223(02)01866-8. PMID 12946886
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] Keane TM, Caddell JM, Taylor KL. Mississippi Scale for Combat-Related Posttraumatic Stress Disorder: three studies in reliability and validity. J Consult Clin Psychol. 1988 Feb;56(1):85-90. doi: 10.1037//0022-006x.56.1.85. No abstract available. PMID 3346454
- [Background] Bovin MJ, Black SK, Rodriguez P, Lunney CA, Kleiman SE, Weathers FW, Schnurr PP, Spira J, Keane TM, Marx BP. Development and validation of a measure of PTSD-related psychosocial functional impairment: The Inventory of Psychosocial Functioning. Psychol Serv. 2018 May;15(2):216-229. doi: 10.1037/ser0000220. PMID 29723024
- [Background] Cyders MA, Littlefield AK, Coffey S, Karyadi KA. Examination of a short English version of the UPPS-P Impulsive Behavior Scale. Addict Behav. 2014 Sep;39(9):1372-6. doi: 10.1016/j.addbeh.2014.02.013. Epub 2014 Mar 3. PMID 24636739
- [Background] Buss AH, Perry M. The aggression questionnaire. J Pers Soc Psychol. 1992 Sep;63(3):452-9. doi: 10.1037//0022-3514.63.3.452. PMID 1403624
- [Background] Monson CM, Schnurr PP, Resick PA, Friedman MJ, Young-Xu Y, Stevens SP. Cognitive processing therapy for veterans with military-related posttraumatic stress disorder. J Consult Clin Psychol. 2006 Oct;74(5):898-907. doi: 10.1037/0022-006X.74.5.898. PMID 17032094
- [Background] Tillman GD, Kimbrell TA, Calley CS, Kraut MA, Freeman TW, Hart J Jr. Repetitive transcranial magnetic stimulation and threat memory: selective reduction of combat threat memory p300 response after right frontal-lobe stimulation. J Neuropsychiatry Clin Neurosci. 2011 Winter;23(1):40-7. doi: 10.1176/jnp.23.1.jnp40. PMID 21304137
- [Background] DeLaRosa BL, Spence JS, Shakal SK, Motes MA, Calley CS, Calley VI, Hart J Jr, Kraut MA. Electrophysiological spatiotemporal dynamics during implicit visual threat processing. Brain Cogn. 2014 Nov;91:54-61. doi: 10.1016/j.bandc.2014.08.003. Epub 2014 Sep 15. PMID 25222294
- [Background] Maguire MJ, Brier MR, Moore PS, Ferree TC, Ray D, Mostofsky S, Hart J Jr, Kraut MA. The influence of perceptual and semantic categorization on inhibitory processing as measured by the N2-P3 response. Brain Cogn. 2009 Dec;71(3):196-203. doi: 10.1016/j.bandc.2009.08.018. Epub 2009 Sep 20. PMID 19773108
- [Background] Calley CS, Motes MA, Chiang HS, Buhl V, Spence JS, Abdi H, Anand R, Maguire M, Estevez L, Briggs R, Freeman T, Kraut MA, Hart J Jr. Threat as a feature in visual semantic object memory. Hum Brain Mapp. 2013 Aug;34(8):1946-55. doi: 10.1002/hbm.22039. Epub 2012 Mar 25. PMID 22451240